CLINICAL TRIAL: NCT01475279
Title: An Open-Label, Multiple-Dose, Single-Center, Sequential, Inpatient Study to Determine the Effect of T89 on Steady-State Pharmacodynamics of Warfarin in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of T89(Dantonic®)on Steady-State Pharmacodynamics of Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: T89-04-US
Record Dates: First submitted 2011-11-14; First posted 2011-11-21 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Warfarin; Dantonic; Pharmacodynamics; Pharmacokinetics; Interaction
MeSH Terms: interventions — Warfarin; T89 herbal drug

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Warfarin; Dantonic — Individual warfarin dose during the study; 225mg Dantonic b.i.d for one week
  Other Names: coumadin

SUMMARY:
The purpose of this study is to evaluate the potential effect of Dantonic on the steady-state pharmacodynamics and pharmacokinetic of warfarin in healthy subjects and safety of the co-administration of Dantonic and warfarin.

DETAILED DESCRIPTION:
Due to a large proportion of patients that could benefit from Dantonic treatment is likely to take warfarin concomitantly. And there is no systematic experience of warfarin drug-drug interaction between Dantonic and warfarin on humans. It is highly relevant to investigate the potential interaction of theses two drugs.

Primary endpoint:

•The change in INR with T89 (Day 25) compared with that without T89 (Day 18)

Secondary endpoints:

* The change in PK variables for R-warfarin and S-warfarin on Day 17 compared with those on Day 24
* Safety assessments across all time points

ELIGIBILITY:
Inclusion Criteria:

1. Nonsmoking male or female with 18-50 years of age and a body mass index (BMI) from 19.0 to 30.0 kg/m2;
2. Healthy adult with no active medical problems or significant chronic diseases as determined by the study doctor based on medical history, physical examination and laboratory evaluations;
3. Taking no medications 2 weeks before Day 0 and during the study, including drugs of abuse, prescription and non prescription medications (including natural health products, Vitamins, and herbals) and did not receive vaccinations;
4. Agree to avoid eating Seville oranges, grapefruits (including grapefruit juice), broccoli, brussels sprouts, charcoal-grilled meats, alcoholic beverages, and caffeine- and theobromine-containing beverages and foods from the time of screening visit and the duration of the study;
5. Agree to maintain adequate birth control, independent from hormonal contraceptive use, from the time of the screening visit and during the study, at the discretion of the investigator;
6. Agree to abstain from alcoholic beverages, caffeinated beverages and orange juice from 6pm the night before a study day until completion of that study day;
7. A negative fecal occult blood test (FOBT) ;
8. Agree to avoid participation in contact sports and/or other activities with significant risk of trauma injury for 7 days after each study day;
9. Subject understands and is willing, able and likely to comply with all study procedures and restrictions;
10. Subject is able to give voluntary oral and written informed consent, at the discretion of the investigator.

Exclusion Criteria:

1. Subjects with an elevated INR (INR> 1.2) at screening visit;
2. No gastrointestinal bleeding history within 12 months prior to screening visit;
3. No history of endoscopically proven peptic ulcer disease;
4. Known hypersensitivity to warfarin;
5. Prosthetic heart valves, mitral stenosis, or other conditions such as recent (<3 months) pulmonary embolism requiring anticoagulant therapy;
6. History or presence of renal and hepatic insufficiency;
7. History of hyperthyroidism;
8. History of any bleeding disorder or hypercoagulation state;
9. Surgical or medical condition liable to interfere with the absorption, metabolism or excretion of warfarin;
10. Regular intake of other medication affecting the process of coagulation or platelet aggregation (during the 2 weeks prior to screening and/or during the run-in and treatment periods);
11. Significant change in diet likely to interfere with the effects of warfarin in the 2 weeks prior to screening and/or during the run-in and treatment periods, at the discretion of the investigator;
12. History of conditions associated with hemorrhagic risk, surgery or head injury within 6 months prior to screening visit;
13. Hematological abnormalities (thrombocytopenia, clinically significant low granulocyte count, anemia, hypofibrinogenaemia, hemophilia, purpura, hemopathy with prolongation of bleeding time);
14. Blood loss/donation >400 mL within 12 weeks prior to the screening visit and/or during the run-in and treatment periods;
15. Known to have serum hepatitis or who are carrier of the hepatitis B surface antigen (HBsAg), or hepatitis C antibody, or have a positive result to the test for HIV antigens and/or antibodies;
16. Pregnancy or lactation;
17. Participation in any other clinical trial or receipt of an investigational drug within 60 days prior to the time of the screening visit, or previous participation in this study;
18. Those subjects unable, in the opinion of the investigator, to comply fully with the trial requirements;
19. Subjects with a recent history (within 24 months prior to the screening visit) of alcoholism or known drug dependence, at the discretion of the investigator;
20. Subjects with positive urine cotinine, urine drug screen and/or alcohol breath test;
21. In the opinion of the investigator, patients with medical history or other factors which may interfere with enrollment or the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The change in INR with T89 (Day 25) compared with that without T89 (Day 18) | outcome measure will be assessed in two weeks and data will be presented up to eight weeks
  The mean INR change with T89 (Day 25) and without T89 (Day 18) will be assessed by standard t test.

SECONDARY OUTCOMES:
The change in PK variables for R-warfarin and S-warfarin on Day 17 compared with those on Day 24 | outcome measure will be assessed in two weeks and data will be presented up to eight weeks
  The S- and R-warfarin concentration time profiles will be listed and displayed graphically. And 90% CI of the geometric mean ratio for Cmax and AUClast of both R- and S-warfarin will be caculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Healthcare Discoveries, LLC d/b/a ICON Development Solutions, San Antonio, Texas, United States